CLINICAL TRIAL: NCT02690922
Title: The Combination of Lower Dosage of Chemotherapy With Tyrosine Kinase Inhibitor to Treat Newly Diagnosed ph+ Acute Lymphoblastic Leukemia Patients
Brief Title: Low-dose Chemotherapy Combine With Tyrosine Kinase Inhibitor to Treat ph+ Acute Lymphoblastic Leukemia Patients
Acronym: TCLDCWTTNDPP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Meng Li, professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJXYXXW
Record Dates: First submitted 2016-01-27; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: ph+ Acute Lymphoblastic Leukemia
MeSH Terms: interventions — Dasatinib; Prednisone; prednylidene; Dexamethasone; Calcium Dobesilate; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ph+ ALL with dasatinib (Experimental): patients in the arm are newly diagnosed ph+ ALL,the patient first receive dexamethasone as pretreatment,then dasatinib and prednisone are used as inductive treatment,and methotrexate to consolidate the therapy.
  Interventions: Drug: Dasatinib; Drug: prednisone; Drug: dexamethasone; Drug: methotrexate

INTERVENTIONS:
Drug: Dasatinib — 100mg (d1-d84)
  Other Names: Sprycel
Drug: prednisone — 60mg/m2 d1-24
  Other Names: Pred
Drug: dexamethasone — 10mg/d 3-7days
  Other Names: Decadron
Drug: methotrexate — 3g/m2 1day
  Other Names: MTX

SUMMARY:
The aim of our study is to improve the major molecular remission(MMR) rate and reduce the cost to treat ph(+) Acute Lymphoblastic Leukemia (ALL) by adjusting chemotherapy regimens and the dosage of Tyrosine Kinase Inhibitor (TKI). lower the classification of chemotherapy drugs, lower the side effect brought by which this would be a grateful news for the patients once this regimens gain a successful result, which is also the final aim of our efforts.

DETAILED DESCRIPTION:
The investigators new therapy regimens: The investigators use dexamethasone 10mg/d(d3-d7) as pre-processing therapy, dasatinib 100mg (d1-d84) plus prednisone 60mg/m2 (d1-24), reduce to d32, as inductive treatment after inductive treatment, if the patient get major molecular remission, patient will get to consolidation therapy, that is methotrexate (MTX) 3g/m2 d1, if not, this patient would be excluded from our trail. after consolidation therapy, if the patient have matched bone marrow donor, the investigators will suggest the patient receipting allogens-stem cell transplantation, otherwise, autogens stem cell transplantation can also be considered once the patient have no applicable bone marrow donor. on the other side, if the patient still not get MMR after this two cycle, maybe the patient can try Car-T, or other chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Get signed the informed consent of patients and family members
2. Age ≥ 18 one full year of life
3. Confirm the ph + ALL at molecular biology level
4. Normal heart and lungs function
5. Normal liver and kidney function

Exclusion Criteria:

1. Leukemia in the nervous system
2. Recurrent patients
3. Allergies associated with any drug in our research
4. At the same time with other organs' malignant tumours
5. participating in other clinical researches at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The rate of major molecular remission after two cycle chemotherapy with MTX and dasatinib | 115 days

SECONDARY OUTCOMES:
Time needed to achieve MMR | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Li Meng, professor, Study Chair — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fujisawa S, Nakamae H, Ogura M, Ishizawa K, Taniwaki M, Utsunomiya A, Matsue K, Takamatsu Y, Usuki K, Tanimoto M, Ishida Y, Akiyama H, Onishi S. Efficacy and safety of dasatinib versus imatinib in Japanese patients with newly diagnosed chronic-phase chronic myeloid leukemia (CML-CP): Subset analysis of the DASISION trial with 2-year follow-up. Int J Hematol. 2014 Feb;99(2):141-53. doi: 10.1007/s12185-013-1470-1. Epub 2013 Dec 20. PMID 24357015
- [Derived] Peng Y, Huang J, Yin J, Meng F, Cao Y, Huang L, Li D, Zhang Y, Zhang D, Meng L, Han Z, Hong Z. Frontline combination of dasatinib and low-intensity chemotherapy in adults with de novo Philadelphia chromosome-positive acute lymphoblastic leukemia. Expert Rev Hematol. 2024 Apr-May;17(4-5):173-180. doi: 10.1080/17474086.2024.2343885. Epub 2024 Apr 24. PMID 38616308